CLINICAL TRIAL: NCT04396730
Title: Cannabidiol and Oral Contraceptive Pills: Exploring a Drug-Drug Interaction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Shaalini Ramanadhan, Clinical Instructor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00020906
Record Dates: First submitted 2020-04-29; First posted 2020-05-21 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Contraception
Keywords: Cannabidiol; Combined oral contraceptives
MeSH Terms: interventions — Cannabidiol; Contraceptives, Oral, Combined

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo followed by cannabidiol (Placebo Comparator): Oral contraceptives will be taken daily for 24 days along with placebo (oral) once daily for cycle 1. During cycle 3, cannabidiol will be taken once daily along with OCPs.
  Interventions: Drug: Cannabidiol Oil; Drug: Placebo; Drug: Combined oral contraceptive pill
- Cannabidiol follow Placebo (Experimental): Oral contraceptives will be taken daily for 24 days along with Cannabidiol 400mg once daily for cycle 1. During cycle 3. placebo will be taken once daily along with OCPs.
  Interventions: Drug: Cannabidiol Oil; Drug: Placebo; Drug: Combined oral contraceptive pill

INTERVENTIONS:
Drug: Cannabidiol Oil — 400 mg Cannabidiol oil will be administered daily along with oral contraceptives daily for 24 days.
  Other Names: Cannabidiol + OCP
Drug: Placebo — Placebo will be administered daily along with oral contraceptives daily for 24 days.
  Other Names: Placebo + OCP
Drug: Combined oral contraceptive pill — All participants will receive oral contraceptives

SUMMARY:
The purpose of this study is to assess how Cannabidiol (CBD) impacts the effectiveness of oral contraceptive (birth control) pills and if CBD changes the possible side effects of birth control pills when CBD and birth control pills are taken at the same time.

This study explores the potential interaction between CBD and birth control pills by assessing serum levels of the contraceptive steroid hormones ethinyl estradiol and levonorgestrel in birth control pill users when they also use CBD.

DETAILED DESCRIPTION:
Participants will be randomized to either the CBD or placebo for cycle one, followed by a washout cycle. For cycle three, participants will take the opposite of what they received in Cycle one. For example if they received CBD during cycle one they will take placebo for cycle 3.

ELIGIBILITY:
Inclusion Criteria:

* Have regular menses (every 21-35 days)
* Not at risk for pregnancy (not sexually active, using a barrier method of birth control, using a copper IUD for birth control, have a partner with a vasectomy, have had a tubal ligation, or in a same sex relationship)
* Generally healthy women between the age of 18 to 35 years old
* English speaking

Exclusion Criteria:

* Active users of hormonal contraception

  1. For combined methods, if they have recently stopped use, they must have had one normal menstrual cycle
  2. For prior Depo-Medroxyprogesterone Acetate users, they must be off of the medication for 2 months and be having regular menstrual cycles
* Pregnancy (less than 6 weeks prior), breastfeeding (less than 6 weeks prior),

  a. If participants have a normal menstrual cycle after these events, they may be considered for enrollment
* Any absolute/relative contraindications to EE and LNG (MEC category 3 or 4 [12]) including impaired liver function, history of deep venous thrombosis, hypertension (> 140/90), diabetes with vascular changes, migraines with aura or neurological changes, history of myocardial infarction, pulmonary embolus, stroke or breast cancer.
* Use of CBD or THC products / Marijuana in the last 30 days
* Use of a known CYP450 inhibitor or inducer (other medication)
* BMI>25
* Metabolic disorders including uncontrolled thyroid dysfunction and Polycystic Ovarian Syndrome
* Impaired liver or renal function
* Smoking/vaping/e-cigarettes
* Prior bariatric surgery
* Decisional impairment
* Incarceration

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration Ethinyl Estradiol | At the end of Cycle 1 (each cycle is 28 days)
  Area under the plasma concentration vs time curve of ethinyl estradiol (EE)
Maximum plasma concentration Ethinyl Estradiol | At the end of Cycle 3 (each cycle is 28 days)
  Area under the plasma concentration vs time curve of ethinyl estradiol (EE)
Maximum plasma concentration of Levonorgestrel | At the end of Cycle 1 (each cycle is 28 days)
  Area under the plasma concentration vs time curve of levonorgestrel (LNG)
Maximum plasma concentration of Levonorgestrel | At the end of Cycle 3 (each cycle is 28 days)
  Area under the plasma concentration vs time curve of levonorgestrel (LNG)

SECONDARY OUTCOMES:
Time to maximum measured plasma concentration (Tmax) | At the end of Cycle 1 (each cycle is 28 days)
  Time to maximum measured plasma concentration of LNG and EE. (Tmax)
Time to maximum measured plasma concentration (Tmax) | At the end of Cycle 3 (each cycle is 28 days)
  Time to maximum measured plasma concentration of LNG and EE. (Tmax)
Time to maximum measured plasma concentration (Cmax) | At the end of Cycle 1 (each cycle is 28 days)
  Time to maximum measured plasma concentration of LNG and EE (Cmax)
Time to maximum measured plasma concentration (Cmax) | At the end of Cycle 3 (each cycle is 28 days)
  Time to maximum measured plasma concentration of LNG and EE (Cmax)
Final time taken for plasma concentration to be reduced by half (t1/2) | At the end of Cycle 1 (each cycle is 28 days)
  Final time taken for plasma concentration of LNG and EE to be reduced by half (t1/2)
Final time taken for plasma concentration to be reduced by half (t1/2) | At the end of Cycle 3 (each cycle is 28 days)
  Final time taken for plasma concentration of LNG and EE to be reduced by half (t1/2)
The area under the plasma concentration of LNG and EE vs. time curve (AUC) | At the end of Cycle 1 (each cycle is 28 days)
  The area under the plasma concentration of LNG and EE vs. time curve (AUC)
The area under the plasma concentration of LNG and EE vs. time curve (AUC) | At the end of Cycle 3 (each cycle is 28 days)
  The area under the plasma concentration of LNG and EE vs. time curve (AUC)
The first-order final elimination rate constant of EE and LNG | At the end of Cycle 1 (each cycle is 28 days)
  The first-order final elimination rate constant of EE and LNG
The first-order final elimination rate constant of EE and LNG | At the end of Cycle 3 (each cycle is 28 days)
  The first-order final elimination rate constant of EE and LNG

CONTACTS AND LOCATIONS:
Overall Officials: Shaalini Ramanadhan, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No